CLINICAL TRIAL: NCT05132712
Title: Effects of Angiotensin Converting Enzyme Inhibitors on Patency of Arterio-Venous Fistulas: A Randomized Controlled Trial
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Armed Forces Post Graduate Medical Institute (AFPGMI), Rawalpindi (Other)
Responsible Party: Principal Investigator, Ayesha Masood, Registrar vascular surgery, Armed Forces Post Graduate Medical Institute (AFPGMI), Rawalpindi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 105471
Record Dates: First submitted 2021-11-22; First posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Vascular Access Complication
MeSH Terms: interventions — Losartan

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Use of ACE inhibitor (Experimental): losartan potassium will be administered 25 mg daily
  Interventions: Drug: Losartan Potassium
- placebo group (Placebo Comparator): matched for age and gender
  Interventions: Drug: multi-vitamins

INTERVENTIONS:
Drug: Losartan Potassium — ACE inhibitor
  Arms: Use of ACE inhibitor
Drug: multi-vitamins — placebo drug
  Arms: placebo group

SUMMARY:
Chronic kidney disease (CKD) is one of the leading health problems imbibing a major portion of health budget worldwide. The global prevalence of CKD is estimated to be 13.4% with approximately 5 to 7 million people needing renal replacement therapy. There is lack of epidemiological surveys regarding CKD but it is estimated to be around 5% and nearly half of them are diabetic. In Pakistan most of the patients undergo hemodialysis as mode of renal replacement as renal transplant centers are few and over burdened. Therefore, a good vascular access for hemodialysis is vital for CKD patients. A functioning arterio-venous fistula (AVF) improves quality of life and morbidity. However, access failure remains a major problem in patients of CKD accounting for third most common cause of admission. There are various options for attaining vascular access but AVF remains the most reliable with less morbidity and better overall patency rate. However, the AVF has its own limitation and has overall patency rate of 50-70% at 1 year and 30-40% at 2 years. This outcome indicates that strategies to prevent occlusion by altering modifiable risk factors are suboptimal and warrant further research.

Patients of CKD often have associated cardiovascular diseases as Ischemic heart disease, left ventricular failure and angina. They are often taking cardio-protective medicines as antiplatelets, angiotensin converting enzymes and calcium channel blockers. Intimal hyperplasia has been shown to be the most important cause of AVF failures.2 Angiotensin II promotes vascular smooth muscle proliferation through various growth factors. Various experimental models have clearly depicted that ACE inhibitors effectively stop smooth muscle growth and intimal hyperplasia in vessel walls. Literature review shows conflicting results in terms of AVF patency when ACE inhibitors are used in conjunction. A study by Jackson RS and colleagues showed that ACE inhibitor were associated with reduced hazard ratio [HR], 0.35; 95% confidence interval [CI], 0.16-0.76; P = .008). Whereas, another study showed no role of ACE inhibitors in preventing graft failure. The possible explanation can be study designs as most studies were retrospective and effects of possible confounders. Moreover, there is lack of research in Pakistan to see the effects of pharmacological drugs on primary patency of AVF among CKD patients.

The rationale of this study is to effectively establish the role of ACE inhibitors in achieving primary patency of AV fistulas while reducing the number of confounders. This will be the first randomized controlled trial conducted in Pakistan. The primary outcome is AVF patency at one year. Secondary outcomes will include graft complications and graft maturation time after surgery.

ELIGIBILITY:
Inclusion Criteria:

All patients who were undergoing Hemodialysis or were intended to start HD within three months between the age of 20 years to 70 years were included in the study

Exclusion Criteria:

* Age less than 20 years or more than 79 years
* In patients who are not expected to start dialysis in next 3 months
* Non-consenting patients
* Patients with diagnosed carcinoma whose life expectancy is less than a year.
* Patients with un-controlled hypertension on multiple regimes of antihypertensive
* Patients allergic to ACE inhibitors

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
primary patency at one year | 1 year

SECONDARY OUTCOMES:
graft complications | 1 year
maturation time of fistula | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Anas Bin Saif, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided